CLINICAL TRIAL: NCT04296630
Title: Utilizing Social Media for Colorectal Cancer Screening: an Innovative Randomized Controlled Trial
Brief Title: Social Media for Colorectal Cancer Screening
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-005
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Cancer Screening
Keywords: Social media; Ad campaigns
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Message #1 (Active Comparator): This arm will receive one of five social media messages that is preferred by our target population through focus groups that are being conducted as part of a previous study.
  Interventions: Other: Social media message #1
- Message #2 (Active Comparator): This arm will receive the second social media message that is preferred by our target population as identified from our previous focus group study.
  Interventions: Other: Social media message #2
- Message #3 (Active Comparator): This arm will receive the third social media message that is preferred by our target population as identified from our previous focus group study.
  Interventions: Other: Social media message #3
- Arm #4 (Active Comparator): This arm will receive the fourth social media message that is preferred by our target population as identified from our previous focus group study.
  Interventions: Other: Social Media Message #4
- Tailored Arm (Active Comparator): This arm will receive social media messages that will be tailored by sex.
  Interventions: Other: Tailored Social Media Message
- Control Arm (No Intervention): This arm will not receive any intervention.

INTERVENTIONS:
Other: Social media message #1 — Social media message promoting colorectal cancer screening
  Arms: Message #1
Other: Social media message #2 — A different social media message promoting colorectal cancer screening
  Arms: Message #2
Other: Social media message #3 — A different social media message promoting colorectal cancer screening
  Arms: Message #3
Other: Social Media Message #4 — A different social media message promoting colorectal cancer screening.
  Arms: Arm #4
Other: Tailored Social Media Message — Tailored social media messages promoting colorectal cancer screening.
  Arms: Tailored Arm

SUMMARY:
Using social media for health promotion is an innovative and emerging approach but remains relatively unexplored in cancer screening. Uptake of colorectal cancer (CRC) screening remains low and standard methods of reaching out are expensive with limited impact. The objective of this study is to conduct a cluster randomized controlled trial (RCT) to test the effectiveness of social media messages for CRC screening on screening intention (primary outcome). The results of this trial will be of interest to Ontario Health and are likely to be taken up by other screening programs looking for innovative and novel ways to increase screening participation. The study results will be easily translatable identifying the most compelling CRC screening messages while the approach can easily be translated to other cancer disease sites with screening programs.

DETAILED DESCRIPTION:
The investigators will conduct a cluster randomized controlled trial (RCT) in Facebook users (aged 50+) in Ontario. Randomization will be done at the level of the forward sortation area (FSA) - the first three characters of the postal code. All FSAs in Ontario will be randomized to one of six study arms - users assigned to each arm will receive one of the social media messages or no message (control). If users click on the message, a webpage with further information on screening will appear and participants will be asked to indicate intention to get screened for CRC. The primary outcome will be intention to screen and secondary outcomes will include other engagement metrics such as reach, cost-per-click, click-through rates, number of likes, number of impressions, and post comments.

This study will inform the feasibility of using social media for CRC screening and identify the most compelling CRC screening messages for the screen-eligible population.

ELIGIBILITY:
Inclusion Criteria:

* Facebook users in Ontario who are between 55-64 years of age

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56000 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening intention | From date of randomization to end of data collection (1 month)
  The proportion of individuals in each arm that click on the ad and confirm their intention to get screened for CRC

SECONDARY OUTCOMES:
Cost-per-click | From date of randomization to end of data collection (1 month)
  The average cost per link click calculated as the total amount spent on the ad campaign divided by total number of link clicks
Click-through-rate | From date of randomization to the end of data collection (1 month)
  Percentage of times that individuals saw the ads and performed a click
Number of likes | At the end of the study period at 1 month
  Total number of Facebook likes for each ad
Number of impressions | At the end of the study period at 1 month
  Number of times that each ad was on screen
Post comments | At the end of the study period at 1 month
  Number of comments on each ad

CONTACTS AND LOCATIONS:
Overall Officials: Nancy N. Baxter, MD, FRCSC, FACS, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to share because the study results will not be at the individual-level and therefore this is not applicable.